CLINICAL TRIAL: NCT02147197
Title: A Randomized, Placebo-Controlled, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of Ulipristal Acetate for the Treatment of Abnormal Uterine Bleeding Associated With Leiomyomas
Brief Title: A Study of the Efficacy and Safety of a 3-month Treatment Course of Ulipristal Acetate for the Treatment of Abnormal Uterine Bleeding Associated With Leiomyomas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UL1309
Record Dates: First submitted 2014-05-21; First posted 2014-05-26 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Leiomyoma; Uterine Hemorrhage
MeSH Terms: conditions — Leiomyoma; Uterine Hemorrhage | interventions — ulipristal acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- UPA 5 mg (Experimental): Ulipristal acetate (UPA) 5 mg tablet plus matching placebo 10 mg tablet, orally, once daily for 12 weeks.
  Interventions: Drug: Ulipristal acetate (UPA); Drug: Placebo
- UPA 10 mg (Experimental): UPA 10 mg tablet plus matching placebo 5 mg tablet, orally, once daily for 12 weeks.
  Interventions: Drug: Ulipristal acetate (UPA); Drug: Placebo
- Placebo (Placebo Comparator): Matching placebo tablets (5 mg and 10 mg), orally, once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ulipristal acetate (UPA) — UPA tablet
  Arms: UPA 10 mg; UPA 5 mg
Drug: Placebo — Matching placebo tablet.

SUMMARY:
This study will evaluate the superiority of ulipristal acetate versus placebo for the treatment of abnormal uterine bleeding associated with uterine fibroids

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal women, 18-50 years, inclusive.
* Cyclic abnormal uterine bleeding (heavy or prolonged).
* Menstrual blood loss (MBL) of ≥ 80 mL as measured by the alkaline hematin method in the first 8 days of menses.
* Minimum of one discrete leiomyoma observable by transvaginal ultrasound.
* Endometrial biopsy without evidence of malignancy or atypical or non-atypical hyperplasia

Exclusion Criteria:

* History of uterine surgery that would interfere with the study endpoints.
* Known coagulation disorder including bleeding disorder or clotting disorder.
* History of, or current uterine, cervix, ovarian, or breast cancer.
* Alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase (ALP), or total bilirubin two times or greater than the upper limit of normal rang

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females with abnormal uterine bleeding associated with leiomyomas were treated in this study.
Enrollment: 157 (Actual)
Dates: Start 2014-03-31 (Actual); Primary Completion 2016-03-29 (Actual); Study Completion 2016-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chan, Study Director — Allergan
Locations (28):
- United States (28):
  - Watson Investigational Site 125, Tucson, Arizona
  - Watson Investigational Site 102, San Diego, California
  - Watson Investigational Site 112, Denver, Colorado
  - Watson Investigational Site 115, Lakewood, Colorado
  - Watson Investigational Site 116, Milford, Connecticut
  - Watson Investigational Site 114, Washington D.C., District of Columbia
  - Watson Investigational Site 106, Clearwater, Florida
  - Watson Investigational Site 122, Lake Worth, Florida
  - Watson Investigational Site 130, Miami, Florida
  - Watson Investigational Site 105, New Port Richey, Florida
  - Watson Investigational Site 104, Orlando, Florida
  - Watson Investigational Site 120, Orlando, Florida
  - Watson Investigational Site 103, Atlanta, Georgia
  - Watson Investigational Site 123, Atlanta, Georgia
  - Watson Investigational Site 111, Augusta, Georgia
  - Watson Investigational Site 124, Idaho Falls, Idaho
  - Watson Investigational Site 131, Brownsburg, Indiana
  - Watson Investigational Site 129, Shawnee Mission, Kansas
  - Watson Investigational Site 132, Metairie, Louisiana
  - Watson Investigational Site 110, Norfolk, Nebraska
  - Watson Investigational Site 113, Albuquerque, New Mexico
  - Watson Investigational Site 121, Raleigh, North Carolina
  - Watson Investigational Site 109, Winston-Salem, North Carolina
  - Watson Investigational Site 107, Columbus, Ohio
  - Watson Investigational Site 119, Jenkintown, Pennsylvania
  - Watson Investigational Site 108, Myrtle Beach, South Carolina
  - Watson Investigational Site 101, Chattanooga, Tennessee
  - Watson Investigational Site 126, Memphis, Tennessee

REFERENCES:
- [Derived] Coyne KS, Harrington A, Currie BM, Chen J, Gillard P, Spies JB. Psychometric validation of the 1-month recall Uterine Fibroid Symptom and Health-Related Quality of Life questionnaire (UFS-QOL). J Patient Rep Outcomes. 2019 Aug 23;3(1):57. doi: 10.1186/s41687-019-0146-x. PMID 31444600
- [Derived] Lukes AS, Soper D, Harrington A, Sniukiene V, Mo Y, Gillard P, Shulman L. Health-Related Quality of Life With Ulipristal Acetate for Treatment of Uterine Leiomyomas: A Randomized Controlled Trial. Obstet Gynecol. 2019 May;133(5):869-878. doi: 10.1097/AOG.0000000000003211. PMID 30969201
- [Derived] Simon JA, Catherino W, Segars JH, Blakesley RE, Chan A, Sniukiene V, Al-Hendy A. Ulipristal Acetate for Treatment of Symptomatic Uterine Leiomyomas: A Randomized Controlled Trial. Obstet Gynecol. 2018 Mar;131(3):431-439. doi: 10.1097/AOG.0000000000002462. PMID 29420395

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching placebo tablet (5 mg and 10 mg), orally, once daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | UPA 5 mg | UPA 10 mg
Started | 56 | 53 | 48
Completed | 47 | 47 | 39
Not Completed | 9 | 6 | 9
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal of Consent | 4 | 3 | 2
Not completed — Lost to Follow-up | 2 | 3 | 1
Not completed — Protocol Violation | 1 | 0 | 3
Not completed — Other Miscellaneous Reasons | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Safety Population consisted of all randomized participants who received at least one dose of study drug.
Groups:
- UPA 5 mg: UPA 5 mg tablet plus matching placebo 10 mg tablet, orally, once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | UPA 5 mg | UPA 10 mg | Total
Number analyzed (Participants) | 56 | 53 | 48 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (5.1) | 40.5 (5.9) | 41.3 (5.1) | 41.1 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 53 | 48 | 157
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Absence of Bleeding During the Last 35 Consecutive Days on Treatment
Description: Participants recorded bleeding in a daily diary. Absence of bleeding was defined as no bleeding days (i.e. no entries for bleeding or heavy bleeding; however, spotting was allowed), during the last 35 consecutive days on treatment in the 12-week Treatment Period.
Time Frame: Last 35 consecutive days on treatment in the 12-week Treatment Period
Population: Intent-to-Treat (ITT) Population included all randomized participants. Data was summarized as per the treatment assigned.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | UPA 5 mg | UPA 10 mg
Number analyzed (Participants) | 56 | 53 | 48
percentage of participants | 1.8 [0.0 to 10.9] | 47.2 [31.6 to 63.2] | 58.3 [41.2 to 74.1]

2. Primary Outcome: Time to Absence of Bleeding on Treatment
Description: Time to absence of bleeding was defined as the duration in days from first dose to the first day in the time interval in which absence of bleeding occurs and persists through the last dose on treatment. The persistence of absence of bleeding occurred for a minimum of 35 consecutive days counting backward from the last dose on treatment in the 12-week Treatment Period.
Time Frame: From first dose up to the end of the 12-week Treatment Period
Population: ITT Population included all randomized participants. Data was summarized as per the treatment assigned.
Measure: Median (97.5% Confidence Interval); unit: days
Arm/Group | Placebo | UPA 5 mg | UPA 10 mg
Number analyzed (Participants) | 56 | 53 | 48
days | NA [NA to NA] — The Median, upper and lower limit of 97.5% Confidence Interval were not estimated due to the low number of participants with events. | NA [6.0 to NA] — The Median and upper limit of 97.5% Confidence Interval were not estimated due to the low number of participants with events. | 9.5 [5.0 to NA] — The upper limit of 97.5% Confidence Interval were not estimated due to the low number of participants with events.

3. Secondary Outcome: Percentage of Participants With Absence of Bleeding From Day 11 Through the End of Treatment
Description: Participants recorded bleeding in a daily diary. Absence of bleeding was defined as no bleeding days (i.e. no entries for bleeding or heavy bleeding; however, spotting was allowed), starting from Day 11 through the end of the 12-week Treatment Period.
Time Frame: Day 11 through the end of the 12-week Treatment Period
Population: ITT Population included all randomized participants. Data was summarized as per the treatment assigned.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | UPA 5 mg | UPA 10 mg
Number analyzed (Participants) | 56 | 53 | 48
percentage of participants | 0.0 [0.0 to 7.5] | 43.4 [28.2 to 59.6] | 58.3 [41.2 to 74.1]

4. Secondary Outcome: Change From Baseline in Uterine Fibroid Symptom and Health-Related Quality of Life Questionnaire (UFS-QOL) Revised Activities Subscale Score at the End of Treatment Period
Description: The UFS-QOL is a uterine fibroid-specific questionnaire consisting of 37 questions developed to evaluate symptoms of uterine fibroids and their impact on health-related quality of life in women with leiomyomas. The first 8 questions comprise the Symptom Severity subscale to assess symptoms experienced by women with uterine leiomyomas, the remaining 29 questions comprise 6 subscales (Concern, Activities, Energy/mood, Control, Self-consciousness, Sexual Function) which overall deal with women's feelings and experiences regarding impact of uterine leiomyoma symptoms on her life. Each item is scored between 1 and 5, where 1=none of the time or not at all and 5=all of the time or a very great deal. A Revised Activities subscale was created to include the most relevant items pertaining to physical and social activities with a total possible score of 0 to 100. Higher Revised Activities subscale scores indicate less impact on activities. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 1-4) to the end of 12-week Treatment Period
Population: Data was summarized as per treatment assigned and included all participants with data at both Baseline and Week 12. The Baseline row shows the actual scores. The results at Week 12 are the difference in scores from Baseline to Week 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UPA 5 mg | UPA 10 mg
Number analyzed (Participants) | 51 | 50 | 43
score on a scale
  Baseline | 34.51 (26.41) | 29.60 (23.34) | 28.15 (23.39)
  Change from Baseline at Week 12 | 18.26 (27.52) | 53.00 (34.36) | 61.04 (31.99)

ADVERSE EVENTS:
Time Frame: From study drug administration until the end of the 12-week off-treatment follow-up period (Up to 24 weeks)
Description: Safety Population consisted of all randomized participants who received at least one dose of study drug.
Arm/Group | Placebo | UPA 5 mg | UPA 10 mg
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/53 | 0/48
Serious Adverse Events (participants affected / at risk) | 1/56 | 1/53 | 2/48
Other Adverse Events (participants affected / at risk) | 4/56 | 8/53 | 12/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=56) | UPA 5 mg (N=53) | UPA 10 mg (N=48)
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=56) | UPA 5 mg (N=53) | UPA 10 mg (N=48)
Hypertension (Vascular disorders) | 0 | 2 | 3
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 3
Hot flush (Vascular disorders) | 0 | 3 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
Nausea (Gastrointestinal disorders) | 3 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.